CLINICAL TRIAL: NCT02323646
Title: A Phase 2, Multi-Center, Parallel Design, Randomized, Double-Blind Study to Evaluate the Safety and Efficacy of 6 and 12 mg Proellex® (Telapristone Acetate) Administered Vaginally in the Treatment of Premenopausal Women With Confirmed Symptomatic Uterine Fibroids
Brief Title: Safety and Efficacy of Telapristone Acetate (Proellex®) Administered Vaginally for the Treatment of Uterine Fibroids
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZPV-201
Record Dates: First submitted 2014-12-18; First posted 2014-12-23 (Estimated); Results first posted 2019-06-14 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Uterine Fibroids
Keywords: uterine fibroids; leiomyoma; fibroid tumor; fibroma
MeSH Terms: conditions — Leiomyoma; Fibroma | interventions — telapristone acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Following the baseline assessment no treatment period, matching placebo, vaginally, once daily for 18 weeks (Course 1) and repeated for an additional 18 weeks (Course 2) following the ODI.
  Interventions: Drug: Placebo
- Telapristone Acetate 6 mg (Experimental): Following the baseline assessment no treatment period, telapristone acetate 6 milligrams (mg), vaginally, once daily for 18 weeks (Course 1) and repeated for an additional 18 weeks (Course 2) following the ODI.
  Interventions: Drug: Telapristone Acetate
- Telapristone Acetate 12 mg (Experimental): Following the baseline assessment no treatment period, telapristone acetate 12mg, vaginally, once daily for 18 weeks (Course 1) and repeated for an additional 18 weeks (Course 2) following the ODI.
  Interventions: Drug: Telapristone Acetate

INTERVENTIONS:
Drug: Placebo — Matching placebo, vaginally, once daily for 18 weeks (Course 1) and repeated for an additional 18 weeks (Course 2) following the ODI.
  Arms: Placebo
Drug: Telapristone Acetate — Telapristone acetate, vaginally, once daily for 18 weeks (Course 1) and repeated for an additional 18 weeks (Course 2) following the ODI.
  Other Names: Proellex®
  Arms: Telapristone Acetate 12 mg; Telapristone Acetate 6 mg

SUMMARY:
The primary objective of this study is to determine the safety and efficacy of two vaginal doses of Proellex® administered for up to 2 courses of treatment (18 weeks each), each separated by an Off-Drug Interval (ODI), to premenopausal women with symptomatic uterine fibroids.

ELIGIBILITY:
Inclusion Criteria:

* Adult females between 18 and 47 years.
* Have a history of at least 3 regular menstrual cycles in which menorrhagia is due to uterine fibroids.
* Must have uterine fibroids.
* Agreement not to attempt to become pregnant during the trial.
* Agreement to use only sanitary pads provided throughout the course of the study, tampon use is prohibited .
* Ability to complete a daily Participant diary and study procedures in compliance with the protocol.
* Have a negative pregnancy test at the Screening and Baseline visits, and subsequent study visits.
* A Body Mass Index (BMI) between 18 and 45 inclusive.
* Menstrual blood loss > 80 milliliters (mL) by alkaline hematin assay.

Exclusion Criteria:

* Post-menopausal woman, defined as either; six (6) months or more (immediately prior to screening visit) without a menstrual period, or prior hysterectomy and/or oophorectomy.
* Pregnant or lactating or is attempting or expecting to become pregnant during the entire study period.
* Received an investigational drug in the 30 days prior to the screening for this study.
* History of Polycystic Ovarian Syndrome (PCOS).
* Concurrent use of any testosterone, progestin, androgen, estrogen, anabolic steroids, Dihydroepiandrosterone (DHEA) or hormonal products for at least 2 weeks prior to screening and during the study.
* Use of oral contraceptives in the preceding 30 days. Use of Depo-Provera® in the preceding 10 months.
* Use of Gonadotropin Releasing Hormone (GnRHas) (e.g. Lupron Depot) within 3 months of the first dose of study drug (Lupron Depot must have a wash-out period of 3 months).
* Has an Intra Uterine device (IUD) in place.
* Known or suspected carcinoma of the breast or reproductive organs.
* Recent history (within past 6 months) of alcoholism or drug abuse.
* Clinically significant abnormal findings on screening examination and laboratory assessments or any condition which in the opinion of the investigator would interfere with the participant's ability to comply with the study instructions or endanger the participant if she took part in the study.

Ages: 18 Years to 47 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2015-02-12 (Actual); Primary Completion 2017-04-06 (Actual); Study Completion 2017-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Chan, Study Director — Allergan
Locations (7):
- United States (7):
  - Fort Lauderdale, Florida
  - Sandy Springs, Georgia
  - Metairie, Louisiana
  - Saginaw, Michigan
  - Raleigh, North Carolina
  - Houston, Texas
  - Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Telapristone Acetate 12 mg: Following the baseline assessment no treatment period, telapristone acetate 12 mg, vaginally, once daily for 18 weeks (Course 1) and repeated for an additional 18 weeks (Course 2) following the ODI.
Period: Treatment Course 1
Arm/Group | Placebo | Telapristone Acetate 6 mg | Telapristone Acetate 12 mg
Started | 14 | 13 | 15
Completed | 11 | 10 | 12
Not Completed | 3 | 3 | 3
Not completed — Adverse Event | 1 | 0 | 1
Not completed — Heavy Bleeding | 1 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2 | 0
Period: Treatment Course 2
Arm/Group | Placebo | Telapristone Acetate 6 mg | Telapristone Acetate 12 mg
Started | 11 | 10 | 12
Completed | 10 | 9 | 9
Not Completed | 1 | 1 | 3
Not completed — Adverse Event | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Non-compliance | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population included all study participants who received at least 1 dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Telapristone Acetate 6 mg | Telapristone Acetate 12 mg | Total
Number analyzed (Participants) | 14 | 13 | 15 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.3 (4.53) | 39.4 (3.55) | 40.9 (3.31) | 40.6 (3.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 15 | 42
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Safety Population included all study participants who received at least 1 dose of study treatment.
  Participants
    Black or African American | 13 | 12 | 14 | 39
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
    White | 1 | 1 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Safety Population included all study participants who received at least 1 dose of study treatment.
  Participants
    Hispanic or Latino | 2 | 1 | 1 | 4
    Not Hispanic or Latino: number analyzed (Participants) | 14 | 13 | 14 | 41
    Not Hispanic or Latino | 12 | 12 | 14 | 38

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants in Amenorrhea at the End of Treatment Course 1
Description: Amenorrhea was defined as any 28-day period during treatment (not including the ODI) without a bleeding intensity score >1. Participants were provided with a daily diary and Pictorial Blood Loss Assessment Chart (PBAC) to record information about the menstrual blood loss (MBL). Bleeding intensity was graded on a 5-point scale where: 1=spotting to 5=heavy bleeding.
Time Frame: At the end of 18-weeks Treatment Course 1
Population: Intent-to-Treat (ITT) population included all participants who were randomized and received study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Telapristone Acetate 6 mg | Telapristone Acetate 12 mg
Number analyzed (Participants) | 14 | 13 | 15
percentage of participants | 0.0 | 53.8 | 46.7
Statistical Analysis 1: Comparison: Placebo vs Telapristone Acetate 6 mg; Test type: Superiority; p = 0.0019, Fisher Exact
Statistical Analysis 2: Comparison: Placebo vs Telapristone Acetate 12 mg; Test type: Superiority; p = 0.0063, Fisher Exact

2. Secondary Outcome: Percentage of Participants in Amenorrhea at the End of Treatment Course 2
Description: Amenorrhea was defined as any 28-day period during treatment (not including the ODI) without a bleeding intensity score >1 after 2 courses of treatment. Participants were provided with a daily diary and (PBAC) to record information about the MBL. Bleeding intensity was graded on a 5-point scale where: 1=spotting to 5=heavy bleeding.
Time Frame: At the end of 18-weeks Treatment Course 2
Population: ITT population included all participants who were randomized and received study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Telapristone Acetate 6 mg | Telapristone Acetate 12 mg
Number analyzed (Participants) | 14 | 13 | 15
percentage of participants | 7.1 | 46.2 | 46.7
Statistical Analysis 1: Comparison: Placebo vs Telapristone Acetate 6 mg; Test type: Superiority; p = 0.0237, Fisher Exact
Statistical Analysis 2: Comparison: Placebo vs Telapristone Acetate 12 mg; Test type: Superiority; p = 0.0272, Fisher Exact

3. Secondary Outcome: Percentage Change in PBAC Scores From Baseline to the End of Treatment Courses 1 and 2
Description: Uterine bleeding was assessed with the use of the PBAC, a validated self-reporting method to estimate menstrual blood loss. Participants recorded daily the number of tampons and towels used and the degree to which individual items were soiled with blood (plus small or large clots). Pictorial scores range from score 1 for slightly stained tampon/towel, 5 for a partially stained tampon/towel, 10 for a completely saturated tampon, 20 for a completely saturated towel, and 5 for each episode of flooding and for each blood clot larger than a quarter in size. Total score can range from 0 (no bleeding) to >500. Higher scores indicate more bleeding. Lower scores indicate less bleeding. A negative change from Baseline indicates improvement (reduction in bleeding).
Time Frame: Baseline (No treatment period) to the end of 18-weeks Treatment Course 1 and the end of 18-weeks Treatment Course 2
Population: ITT population included all participants who were randomized and received study drug. Number analyzed is the number of participants with data available at the given time-point.
Measure: Mean (Standard Deviation); unit: percentage change in PBAC score
Arm/Group | Placebo | Telapristone Acetate 6 mg | Telapristone Acetate 12 mg
Number analyzed (Participants) | 14 | 13 | 15
percentage change in PBAC score
  Percentage Change from BL: Course 1 | -1.21 (100.850) | -55.43 (87.522) | -43.85 (82.634)
  Percentage Change from BL: Course 2: number analyzed (Participants) | 11 | 10 | 12
  Percentage Change from BL: Course 2 | -43.52 (37.967) | -91.02 (18.367) | -77.42 (34.762)
Statistical Analysis 1: Comparison: Placebo vs Telapristone Acetate 6 mg; Percentage change in the last value on drug Course 1; Test type: Superiority; p = 0.0145, Wilcoxon Rank-Sum Test
Statistical Analysis 2: Comparison: Placebo vs Telapristone Acetate 12 mg; Percentage change in the last value on drug Course 1; Test type: Superiority; p = 0.0662, Wilcoxon Rank-Sum Test
Statistical Analysis 3: Comparison: Placebo vs Telapristone Acetate 6 mg; Percentage change in the last value on drug Course 2; Test type: Superiority; p = 0.0061, Wilcoxon Rank-Sum Test
Statistical Analysis 4: Comparison: Placebo vs Telapristone Acetate 12 mg; Percentage change in the last value on drug Course 2; Test type: Superiority; p = 0.0296, Wilcoxon Rank-Sum Test

4. Secondary Outcome: Percentage Change in Transformed Total Uterine Fibroid System Quality of Life Survey System Severity (UFS-SSS) Score From Baseline to the End of Treatment Courses 1 and 2 and the Course 2 Week 24 Follow-up Visit
Description: UFS-SSS is an 8 question assessment tool used to measure symptom severity and has been validated as a three month look back questionnaire. Each question was answered on a 5-point scale where 1=Not at all to 5=A very great deal. The sum of the total scores was transformed to a range of 0=no symptoms (best) to 100=most severe symptoms (worst). A negative percentage change from Baseline indicates improvement.
Time Frame: Baseline (No treatment period) to the end of 18-weeks Treatment Course 1, the end of 18-weeks Treatment Course 2 and the Course 2 Week 24 Follow-up Visit
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage change in UFS-SSS score
Arm/Group | Placebo | Telapristone Acetate 6 mg | Telapristone Acetate 12 mg
Number analyzed (Participants) | 14 | 13 | 15
percentage change in UFS-SSS score
  Percentage Change from BL: Course 1 | -33.54 (30.981) | -49.68 (37.927) | -42.27 (45.842)
  Percentage Change from BL: Course 2: number analyzed (Participants) | 11 | 10 | 12
  Percentage Change from BL: Course 2 | -31.11 (33.577) | -43.69 (35.919) | -37.98 (46.287)
  Percentage Change: Course 2, Week 24 Follow-up: number analyzed (Participants) | 9 | 9 | 9
  Percentage Change: Course 2, Week 24 Follow-up | -37.38 (30.153) | -26.90 (26.126) | -14.66 (41.842)
Statistical Analysis 1: Comparison: Placebo vs Telapristone Acetate 6 mg; Percentage Change from BL: Course 1; Test type: Superiority; p = 0.2642, Wilcoxon Rank-Sum Test
Statistical Analysis 2: Comparison: Placebo vs Telapristone Acetate 12 mg; Percentage Change from BL: Course 1; Test type: Superiority; p = 0.4383, Wilcoxon Rank-Sum Test
Statistical Analysis 3: Comparison: Placebo vs Telapristone Acetate 6 mg; Percentage Change from BL: Course 2; Test type: Superiority; p = 0.5333, Wilcoxon Rank-Sum Test
Statistical Analysis 4: Comparison: Placebo vs Telapristone Acetate 12 mg; Percentage Change from BL: Course 2; Test type: Superiority; p = 0.8791, Wilcoxon Rank-Sum Test
Statistical Analysis 5: Comparison: Placebo vs Telapristone Acetate 6 mg; Percentage Change: Course 2, Week 24 Follow-up; Test type: Superiority; p = 0.3666, Wilcoxon Rank-Sum Test
Statistical Analysis 6: Comparison: Placebo vs Telapristone Acetate 12 mg; Percentage Change: Course 2, Week 24 Follow-up; Test type: Superiority; p = 0.3450, Wilcoxon Rank-Sum Test

5. Secondary Outcome: Percentage Change in the Individual UFS-SSS Subscale Score Question 1 From Baseline to the End of Treatment Courses 1 and 2 and the Course 2 Week 24 Follow-up Visit
Description: UFS-SSS is an 8 question assessment tool used to measure symptom severity and has been validated as a three month look back questionnaire. The participant answered UFS-SSS subscale question 1: During the previous 3 months how distressed were you by "heavy bleeding during your menstrual period"? using a 5-point scale where 1=Not at all to 5=A very great deal. A negative percentage change from Baseline indicates improvement.
Time Frame: as for outcome 4
Population: ITT population consisted of all participants who were randomized and received study drug. Number analyzed is the number of participants with data available at the given time-point.
Measure: Mean (Standard Deviation); unit: percentage change in UFS-SSS score
Arm/Group | Placebo | Telapristone Acetate 6 mg | Telapristone Acetate 12 mg
Number analyzed (Participants) | 14 | 13 | 15
percentage change in UFS-SSS score
  Percentage Change from BL: Course 1: number analyzed (Participants) | 12 | 12 | 12
  Percentage Change from BL: Course 1 | -19.58 (27.672) | -52.50 (33.811) | -53.75 (28.052)
  Percentage Change from BL: Course 2: number analyzed (Participants) | 10 | 10 | 10
  Percentage Change from BL: Course 2 | -21.00 (30.074) | -55.00 (34.319) | -60.50 (27.330)
  Percentage Change: Course 2, Week 24 Follow-up: number analyzed (Participants) | 9 | 9 | 9
  Percentage Change: Course 2, Week 24 Follow-up | -31.67 (41.003) | -23.89 (31.798) | -22.22 (26.471)
Statistical Analysis 1: Comparison: Placebo vs Telapristone Acetate 6 mg; Percentage Change from BL: Course 1; Test type: Superiority; p = 0.0473, Wilcoxon Rank-Sum Test
Statistical Analysis 2: Comparison: Placebo vs Telapristone Acetate 12 mg; Percentage Change from BL: Course 1; Test type: Superiority; p = 0.0191, Wilcoxon Rank-Sum Test
Statistical Analysis 3: Comparison: Placebo vs Telapristone Acetate 6 mg; Percentage Change from BL: Course 2; Test type: Superiority; p = 0.0749, Wilcoxon Rank-Sum Test
Statistical Analysis 4: Comparison: Placebo vs Telapristone Acetate 12 mg; Percentage Change from BL: Course 2; Test type: Superiority; p = 0.0233, Wilcoxon Rank-Sum Test
Statistical Analysis 5: Comparison: Placebo vs Telapristone Acetate 6 mg; Percentage Change from BL: Course 2, Week 24 Follow-up Visit; Test type: Superiority; p = 0.7569, Wilcoxon Rank-Sum Test
Statistical Analysis 6: Comparison: Placebo vs Telapristone Acetate 12 mg; Percentage Change from BL: Course 2, Week 24 Follow-up Visit; Test type: Superiority; p = 0.5399, Wilcoxon Rank-Sum Test

6. Secondary Outcome: Percentage Change in the Individual UFS-SSS Subscale Score Question 2 From Baseline to the End of Treatment Courses 1 and 2 and the Course 2 Week 24 Follow-up Visit
Description: UFS-SSS is an 8 question assessment tool used to measure symptom severity and has been validated as a three month look back questionnaire. The participant answered UFS-SSS subscale question 2: During the previous 3 months how distressed were you by "passing blood clots during your menstrual period"? using a 5-point scale where 1=Not at all to 5=A very great deal. A negative percentage change from Baseline indicates improvement.
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percentage change in UFS-SSS score
Arm/Group | Placebo | Telapristone Acetate 6 mg | Telapristone Acetate 12 mg
Number analyzed (Participants) | 14 | 13 | 15
percentage change in UFS-SSS score
  Percentage Change from BL: Course 1: number analyzed (Participants) | 12 | 12 | 12
  Percentage Change from BL: Course 1 | -34.03 (28.431) | -49.03 (36.205) | -21.81 (108.137)
  Percentage Change from BL: Course 2: number analyzed (Participants) | 10 | 10 | 10
  Percentage Change from BL: Course 2 | -30.67 (26.646) | -43.83 (40.484) | -45.00 (57.542)
  Percentage Change: Course 2, Week 24 Follow-up: number analyzed (Participants) | 9 | 9 | 9
  Percentage Change: Course 2, Week 24 Follow-up | -45.00 (29.686) | 6.85 (47.232) | 2.78 (116.916)
Statistical Analysis 1: Comparison: Placebo vs Telapristone Acetate 6 mg; Percentage Change from BL: Course 1; Test type: Superiority; p = 0.1683, Wilcoxon Rank-Sum Test
Statistical Analysis 2: Comparison: Placebo vs Telapristone Acetate 12 mg; Percentage Change from BL: Course 1; Test type: Superiority; p = 0.2560, Wilcoxon Rank-Sum Test
Statistical Analysis 3: Comparison: Placebo vs Telapristone Acetate 6 mg; Percentage Change from BL: Course 2; Test type: Superiority; p = 0.4997, Wilcoxon Rank-Sum Test
Statistical Analysis 4: Comparison: Placebo vs Telapristone Acetate 12 mg; Percentage Change from BL: Course 2; Test type: Superiority; p = 0.1334, Wilcoxon Rank-Sum Test
Statistical Analysis 5: Comparison: Placebo vs Telapristone Acetate 6 mg; Percentage Change from BL: Course 2, Week 24 Follow-up Visit; Test type: Superiority; p = 0.0323, Wilcoxon Rank-Sum Test
Statistical Analysis 6: Comparison: Placebo vs Telapristone Acetate 12 mg; Percentage Change from BL: Course 2, Week 24 Follow-up Visit; Test type: Superiority; p = 0.3847, Wilcoxon Rank-Sum Test

7. Secondary Outcome: Percentage Change in the Individual UFS-SSS Subscale Score Question 3 From Baseline to the End of Treatment Courses 1 and 2 and the Course 2 Week 24 Follow-up Visit
Description: UFS-SSS is an 8 question assessment tool used to measure symptom severity and has been validated as a three month look back questionnaire. The participant answered UFS-SSS subscale question 3: During the previous 3 months how distressed were you by "fluctuation in the duration of your menstrual period compared to your previous cycle"? using a 5-point scale where 1=Not at all to 5=A very great deal. A negative percentage change from Baseline indicates improvement.
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percentage change in UFS-SSS score
Arm/Group | Placebo | Telapristone Acetate 6 mg | Telapristone Acetate 12 mg
Number analyzed (Participants) | 14 | 13 | 15
percentage change in UFS-SSS score
  Percentage Change from BL: Course 1: number analyzed (Participants) | 12 | 12 | 12
  Percentage Change from BL: Course 1 | -16.39 (26.178) | -26.81 (37.176) | 21.94 (109.882)
  Percentage Change from BL: Course 2: number analyzed (Participants) | 10 | 10 | 10
  Percentage Change from BL: Course 2 | 38.67 (135.664) | -19.33 (55.729) | -21.67 (48.305)
  Percentage Change: Course 2, Week 24 Follow-up: number analyzed (Participants) | 9 | 9 | 9
  Percentage Change: Course 2, Week 24 Follow-up | 3.70 (62.086) | 14.44 (37.118) | 20.00 (45.826)
Statistical Analysis 1: Comparison: Placebo vs Telapristone Acetate 6 mg; Percentage Change from BL: Course 1; Test type: Superiority; p = 0.6356, Wilcoxon Rank-Sum Test
Statistical Analysis 2: Comparison: Placebo vs Telapristone Acetate 12 mg; Percentage Change from BL: Course 1; Test type: Superiority; p = 0.9539, Wilcoxon Rank-Sum Test
Statistical Analysis 3: Comparison: Placebo vs Telapristone Acetate 6 mg; Percentage Change from BL: Course 2; Test type: Superiority; p = 0.5219, Wilcoxon Rank-Sum Test
Statistical Analysis 4: Comparison: Placebo vs Telapristone Acetate 12 mg; Percentage Change from BL: Course 2; Test type: Superiority; p = 0.2678, Wilcoxon Rank-Sum Test
Statistical Analysis 5: Comparison: Placebo vs Telapristone Acetate 6 mg; Percentage Change from BL: Course 2, Week 24 Follow-up Visit; Test type: Superiority; p = 0.3086, Wilcoxon Rank-Sum Test
Statistical Analysis 6: Comparison: Placebo vs Telapristone Acetate 12 mg; Percentage Change from BL: Course 2, Week 24 Follow-up Visit; Test type: Superiority; p = 0.3847, Wilcoxon Rank-Sum Test

8. Secondary Outcome: Percentage Change in the Individual UFS-SSS Subscale Score Question 4 From Baseline to the End of Treatment Courses 1 and 2 and the Course 2 Week 24 Follow-up Visit
Description: UFS-SSS is an 8 question assessment tool used to measure symptom severity and has been validated as a three month look back questionnaire. The participant answered UFS-SSS subscale question 4: During the previous 3 months how distressed were you by "fluctuation in the length of your monthly cycle compared to your previous cycles"? using a 5-point scale where 1=Not at all to 5=A very great deal. A negative percentage change from Baseline indicates improvement.
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percentage change in UFS-SSS score
Arm/Group | Placebo | Telapristone Acetate 6 mg | Telapristone Acetate 12 mg
Number analyzed (Participants) | 14 | 13 | 15
percentage change in UFS-SSS score
  Percentage Change from BL: Course 1: number analyzed (Participants) | 12 | 12 | 12
  Percentage Change from BL: Course 1 | -29.31 (25.785) | -19.44 (65.452) | 65.28 (136.090)
  Percentage Change from BL: Course 2: number analyzed (Participants) | 10 | 10 | 10
  Percentage Change from BL: Course 2 | 10.17 (45.443) | -40.50 (35.677) | 51.67 (165.216)
  Percentage Change: Course 2, Week 24 Follow-up: number analyzed (Participants) | 9 | 9 | 9
  Percentage Change: Course 2, Week 24 Follow-up | 12.22 (84.967) | -17.41 (38.838) | 97.22 (120.185)
Statistical Analysis 1: Comparison: Placebo vs Telapristone Acetate 6 mg; Percentage Change from BL: Course 1; Test type: Superiority; p = 0.8393, Wilcoxon Rank-Sum Test
Statistical Analysis 2: Comparison: Placebo vs Telapristone Acetate 12 mg; Percentage Change from BL: Course 1; Test type: Superiority; p = 0.1361, Wilcoxon Rank-Sum Test
Statistical Analysis 3: Comparison: Placebo vs Telapristone Acetate 6 mg; Percentage Change from BL: Course 2; Test type: Superiority; p = 0.0382, Wilcoxon Rank-Sum Test
Statistical Analysis 4: Comparison: Placebo vs Telapristone Acetate 12 mg; Percentage Change from BL: Course 2; Test type: Superiority; p = 0.6273, Wilcoxon Rank-Sum Test
Statistical Analysis 5: Comparison: Placebo vs Telapristone Acetate 6 mg; Percentage Change from BL: Course 2, Week 24 Follow-up Visit; Test type: Superiority; p = 0.8237, Wilcoxon Rank-Sum Test
Statistical Analysis 6: Comparison: Placebo vs Telapristone Acetate 12 mg; Percentage Change from BL: Course 2, Week 24 Follow-up Visit; Test type: Superiority; p = 0.1370, Wilcoxon Rank-Sum Test

9. Secondary Outcome: Percentage Change in the Individual UFS-SSS Subscale Score Question 5 From Baseline to the End of Treatment Courses 1 and 2 and the Course 2 Week 24 Follow-up Visit
Description: UFS-SSS is an 8 question assessment tool used to measure symptom severity and has been validated as a three month look back questionnaire. The participant answered UFS-SSS subscale question 5: During the previous 3 months how distressed were you by "feeling tightness or pressure in your pelvic area"? using a 5-point scale where 1=Not at all to 5=A very great deal. A negative percentage change from Baseline indicates improvement.
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percentage change in UFS-SSS score
Arm/Group | Placebo | Telapristone Acetate 6 mg | Telapristone Acetate 12 mg
Number analyzed (Participants) | 14 | 13 | 15
percentage change in UFS-SSS score
  Percentage Change from BL: Course 1: number analyzed (Participants) | 12 | 12 | 12
  Percentage Change from BL: Course 1 | -33.61 (36.054) | -41.11 (30.939) | -53.33 (27.220)
  Percentage Change from BL: Course 2: number analyzed (Participants) | 10 | 10 | 10
  Percentage Change from BL: Course 2 | -33.83 (29.419) | -36.83 (36.847) | -10.67 (57.811)
  Percentage Change: Course 2, Week 24 Follow-up: number analyzed (Participants) | 9 | 9 | 9
  Percentage Change: Course 2, Week 24 Follow-up | -27.22 (42.76) | -7.04 (49.137) | 0.37 (66.378)
Statistical Analysis 1: Comparison: Placebo vs Telapristone Acetate 6 mg; Percentage Change from BL: Course 1; Test type: Superiority; p = 0.7949, Wilcoxon Rank-Sum Test
Statistical Analysis 2: Comparison: Placebo vs Telapristone Acetate 12 mg; Percentage Change from BL: Course 1; Test type: Superiority; p = 0.1928, Wilcoxon Rank-Sum Test
Statistical Analysis 3: Comparison: Placebo vs Telapristone Acetate 6 mg; Percentage Change from BL: Course 2; Test type: Superiority; p = 1.0000, Wilcoxon Rank-Sum Test
Statistical Analysis 4: Comparison: Placebo vs Telapristone Acetate 12 mg; Percentage Change from BL: Course 2; Test type: Superiority; p = 0.3920, Wilcoxon Rank-Sum Test
Statistical Analysis 5: Comparison: Placebo vs Telapristone Acetate 6 mg; Percentage Change from BL: Course 2, Week 24 Follow-up Visit; Test type: Superiority; p = 0.5410, Wilcoxon Rank-Sum Test
Statistical Analysis 6: Comparison: Placebo vs Telapristone Acetate 12 mg; Percentage Change from BL: Course 2, Week 24 Follow-up Visit; Test type: Superiority; p = 0.4602, Wilcoxon Rank-Sum Test

10. Secondary Outcome: Percentage Change in the Individual UFS-SSS Subscale Score Question 6 From Baseline to the End of Treatment Courses 1 and 2 and the Course 2 Week 24 Follow-up Visit
Description: UFS-SSS is an 8 question assessment tool used to measure symptom severity and has been validated as a three month look back questionnaire. The participant answered UFS-SSS subscale question 6: During the previous 3 months how distressed were you by "frequent urination during the daytime hours"? using a 5-point scale where 1=Not at all to 5=A very great deal. A negative percentage change from Baseline indicates improvement.
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percentage change in UFS-SSS score
Arm/Group | Placebo | Telapristone Acetate 6 mg | Telapristone Acetate 12 mg
Number analyzed (Participants) | 14 | 13 | 15
percentage change in UFS-SSS score
  Percentage Change from BL: Course 1: number analyzed (Participants) | 12 | 12 | 12
  Percentage Change from BL: Course 1 | -19.72 (32.943) | -25.97 (24.365) | -40.28 (26.235)
  Percentage Change from BL: Course 2: number analyzed (Participants) | 10 | 10 | 10
  Percentage Change from BL: Course 2 | -30.83 (29.400) | -27.50 (32.272) | -25.67 (50.511)
  Percentage Change: Course 2, Week 24 Follow-up: number analyzed (Participants) | 9 | 9 | 9
  Percentage Change: Course 2, Week 24 Follow-up | -17.59 (35.080) | -8.15 (35.711) | -17.41 (35.080)
Statistical Analysis 1: Comparison: Placebo vs Telapristone Acetate 6 mg; Percentage Change from BL: Course 1; Test type: Superiority; p = 0.9536, Wilcoxon Rank-Sum Test
Statistical Analysis 2: Comparison: Placebo vs Telapristone Acetate 12 mg; Percentage Change from BL: Course 1; Test type: Superiority; p = 0.1355, Wilcoxon Rank-Sum Test
Statistical Analysis 3: Comparison: Placebo vs Telapristone Acetate 6 mg; Percentage Change from BL: Course 2; Test type: Superiority; p = 0.9396, Wilcoxon Rank-Sum Test
Statistical Analysis 4: Comparison: Placebo vs Telapristone Acetate 12 mg; Percentage Change from BL: Course 2; Test type: Superiority; p = 0.9102, Wilcoxon Rank-Sum Test
Statistical Analysis 5: Comparison: Placebo vs Telapristone Acetate 6 mg; Percentage Change from BL: Course 2, Week 24 Follow-up Visit; Test type: Superiority; p = 0.6266, Wilcoxon Rank-Sum Test
Statistical Analysis 6: Comparison: Placebo vs Telapristone Acetate 12 mg; Percentage Change from BL: Course 2, Week 24 Follow-up Visit; Test type: Superiority; p = 0.9302, Wilcoxon Rank-Sum Test

11. Secondary Outcome: Percentage Change in the Individual UFS-SSS Subscale Score Question 7 From Baseline to the End of Treatment Courses 1 and 2 and the Course 2 Week 24 Follow-up Visit
Description: UFS-SSS is an 8 question assessment tool used to measure symptom severity and has been validated as a three month look back questionnaire. The participant answered UFS-SSS subscale question 7: During the previous 3 months how distressed were you by "frequent nighttime urination"? using a 5-point scale where 1=Not at all to 5=A very great deal. A negative percentage change from Baseline indicates improvement.
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percentage change in UFS-SSS score
Arm/Group | Placebo | Telapristone Acetate 6 mg | Telapristone Acetate 12 mg
Number analyzed (Participants) | 14 | 13 | 15
percentage change in UFS-SSS score
  Percentage Change from BL: Course 1: number analyzed (Participants) | 12 | 12 | 12
  Percentage Change from BL: Course 1 | -30.83 (26.443) | -29.03 (32.539) | -30.69 (41.209)
  Percentage Change from BL: Course 2: number analyzed (Participants) | 10 | 10 | 10
  Percentage Change from BL: Course 2 | -31.83 (29.819) | -45.17 (24.999) | -7.67 (59.277)
  Percentage Change: Course 2, Week 24 Follow-up: number analyzed (Participants) | 9 | 9 | 9
  Percentage Change: Course 2, Week 24 Follow-up | -36.30 (24.463) | -33.15 (20.008) | -27.59 (39.678)
Statistical Analysis 1: Comparison: Placebo vs Telapristone Acetate 6 mg; Percentage Change from BL: Course 1; Test type: Superiority; p = 0.8170, Wilcoxon Rank-Sum Test
Statistical Analysis 2: Comparison: Placebo vs Telapristone Acetate 12 mg; Percentage Change from BL: Course 1; Test type: Superiority; p = 0.8177, Wilcoxon Rank-Sum Test
Statistical Analysis 3: Comparison: Placebo vs Telapristone Acetate 6 mg; Percentage Change from BL: Course 2; Test type: Superiority; p = 0.3167, Wilcoxon Rank-Sum Test
Statistical Analysis 4: Comparison: Placebo vs Telapristone Acetate 12 mg; Percentage Change from BL: Course 2; Test type: Superiority; p = 0.5503, Wilcoxon Rank-Sum Test
Statistical Analysis 5: Comparison: Placebo vs Telapristone Acetate 6 mg; Percentage Change from BL: Course 2, Week 24 Follow-up Visit; Test type: Superiority; p = 0.6929, Wilcoxon Rank-Sum Test
Statistical Analysis 6: Comparison: Placebo vs Telapristone Acetate 12 mg; Percentage Change from BL: Course 2, Week 24 Follow-up Visit; Test type: Superiority; p = 0.7260, Wilcoxon Rank-Sum Test

12. Secondary Outcome: Percentage Change in the Individual UFS-SSS Subscale Score Question 8 From Baseline to the End of Treatment Courses 1 and 2 and the Course 2 Week 24 Follow-up Visit
Description: UFS-SSS is an 8 question assessment tool used to measure symptom severity and has been validated as a three month look back questionnaire. The participant answered UFS-SSS subscale question 8: During the previous 3 months how distressed were you by "feeling fatigued"? using a 5-point scale where 1=Not at all to 5=A very great deal. A negative percentage change from Baseline indicates improvement.
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percentage change in UFS-SSS score
Arm/Group | Placebo | Telapristone Acetate 6 mg | Telapristone Acetate 12 mg
Number analyzed (Participants) | 14 | 13 | 15
percentage change in UFS-SSS score
  Percentage Change from BL: Course 1: number analyzed (Participants) | 12 | 12 | 12
  Percentage Change from BL: Course 1 | -30.42 (27.174) | -40.69 (29.759) | -38.33 (65.308)
  Percentage Change from BL: Course 2: number analyzed (Participants) | 10 | 10 | 10
  Percentage Change from BL: Course 2 | -28.33 (25.784) | -32.33 (28.976) | -27.50 (37.509)
  Percentage Change: Course 2, Week 24 Follow-up: number analyzed (Participants) | 9 | 9 | 9
  Percentage Change: Course 2, Week 24 Follow-up | -27.59 (27.299) | -22.59 (19.421) | -12.22 (29.059)
Statistical Analysis 1: Comparison: Placebo vs Telapristone Acetate 6 mg; Percentage Change from BL: Course 1; Test type: Superiority; p = 0.3896, Wilcoxon Rank-Sum Test
Statistical Analysis 2: Comparison: Placebo vs Telapristone Acetate 12 mg; Percentage Change from BL: Course 1; Test type: Superiority; p = 0.1358, Wilcoxon Rank-Sum Test
Statistical Analysis 3: Comparison: Placebo vs Telapristone Acetate 6 mg; Percentage Change from BL: Course 2; Test type: Superiority; p = 0.7903, Wilcoxon Rank-Sum Test
Statistical Analysis 4: Comparison: Placebo vs Telapristone Acetate 12 mg; Percentage Change from BL: Course 2; Test type: Superiority; p = 0.8206, Wilcoxon Rank-Sum Test
Statistical Analysis 5: Comparison: Placebo vs Telapristone Acetate 6 mg; Percentage Change from BL: Course 2, Week 24 Follow-up Visit; Test type: Superiority; p = 0.7891, Wilcoxon Rank-Sum Test
Statistical Analysis 6: Comparison: Placebo vs Telapristone Acetate 12 mg; Percentage Change from BL: Course 2, Week 24 Follow-up Visit; Test type: Superiority; p = 0.4010, Wilcoxon Rank-Sum Test

13. Secondary Outcome: Percentage Change in Total Uterine Fibroid Volume From Baseline to the End of Treatment Courses 1 and 2
Description: The total uterine fibroid volume was measured by Magnetic Resonance Imaging (MRI). A negative change from Baseline indicates improvement.
Time Frame: Baseline (No treatment period) to the end of 18-weeks Treatment Course 1 and the end of 18-weeks Treatment Course 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage change in fibroid volume
Arm/Group | Placebo | Telapristone Acetate 6 mg | Telapristone Acetate 12 mg
Number analyzed (Participants) | 14 | 13 | 15
percentage change in fibroid volume
  Percentage Change from BL: Course 1 | 1.41 (31.115) | -28.26 (26.705) | -13.84 (29.167)
  Percentage Change from BL: Course 2: number analyzed (Participants) | 11 | 10 | 12
  Percentage Change from BL: Course 2 | -3.72 (31.316) | -36.39 (40.892) | -13.06 (42.234)
Statistical Analysis 1: Comparison: Placebo vs Telapristone Acetate 6 mg; Percentage Change from BL: Course 1; Test type: Superiority; p = 0.0294, Wilcoxon Rank-Sum Test
Statistical Analysis 2: Comparison: Placebo vs Telapristone Acetate 12 mg; Percentage Change from BL: Course 1; Test type: Superiority; p = 0.1934, Wilcoxon Rank-Sum Test
Statistical Analysis 3: Comparison: Placebo vs Telapristone Acetate 6 mg; Percentage Change from BL: Course 2; Test type: Superiority; p = 0.0442, Wilcoxon Rank-Sum Test
Statistical Analysis 4: Comparison: Placebo vs Telapristone Acetate 12 mg; Percentage Change from BL: Course 2; Test type: Superiority; p = 0.8314, Wilcoxon Rank-Sum Test

ADVERSE EVENTS:
Time Frame: From first dose of study drug through 30 days after the last dose of study drug (approximately 46 weeks)
Description: Safety Population included all study participants who received at least 1 dose of study treatment.
Arm/Group | Placebo | Telapristone Acetate 6 mg | Telapristone Acetate 12 mg
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/13 | 0/15
Serious Adverse Events (participants affected / at risk) | 2/14 | 2/13 | 2/15
Other Adverse Events (participants affected / at risk) | 13/14 | 13/13 | 11/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=14) | Telapristone Acetate 6 mg (N=13) | Telapristone Acetate 12 mg (N=15)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Chest injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Alcoholism (Psychiatric disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=14) | Telapristone Acetate 6 mg (N=13) | Telapristone Acetate 12 mg (N=15)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0
Type 2 diabetes mellitus (Endocrine disorders) | 1 | 0 | 0
Glaucoma (Eye disorders) | 1 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 0
Catheter site inflammation (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 2
Hot flush (General disorders) | 1 | 2 | 1
Influenza like illness (General disorders) | 1 | 0 | 1
Metaplasia (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 2
Asthma (Immune system disorders) | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 1
Bacterial vaginosis (Infections and infestations) | 2 | 0 | 0
Cystitis (Infections and infestations) | 1 | 1 | 0
Fungal infection (Infections and infestations) | 1 | 2 | 0
Fungal skin infection (Infections and infestations) | 1 | 0 | 0
Pelvic inflammatory disease (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0 | 2
Vulvovaginitis trichomonal (Infections and infestations) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood glucose increased (Investigations) | 0 | 1 | 0
Blood pressure increased (Investigations) | 1 | 1 | 1
Bone density decreased (Investigations) | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 1
Smear cervix abnormal (Investigations) | 1 | 0 | 0
Weight increased (Investigations) | 1 | 1 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 2 | 1
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Breast tenderness (Reproductive system and breast disorders) | 0 | 0 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 1 | 3
Dysmenorrhoea (Reproductive system and breast disorders) | 2 | 0 | 1
Endometrial hypertrophy (Reproductive system and breast disorders) | 2 | 5 | 6
Genital rash (Reproductive system and breast disorders) | 0 | 1 | 0
Libido increased (Reproductive system and breast disorders) | 0 | 1 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1 | 2
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1
Vaginal infection (Reproductive system and breast disorders) | 1 | 0 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 1 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus genital (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dizziness (Vascular disorders) | 1 | 1 | 2
Hypertension (Vascular disorders) | 1 | 1 | 1
Migraine (Vascular disorders) | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review.The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2016-06-20): https://cdn.clinicaltrials.gov/large-docs/46/NCT02323646/Prot_000.pdf
  • Statistical Analysis Plan (2016-04-06): https://cdn.clinicaltrials.gov/large-docs/46/NCT02323646/SAP_001.pdf